CLINICAL TRIAL: NCT05963893
Title: Cooperative Planning Process With the University Community to Sit Less, Move More and Improve Mental Health Though a Gendered Enviromental Approach: the Uni4Move Project
Brief Title: Promoting a Healthy Life Through Gender Equity
Acronym: Uni4Move
Status: Not yet recruiting | Type: Observational
Sponsor: Fundació Universitària del Bages (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_14_PRI
Record Dates: First submitted 2023-07-05; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Mental Health Wellness 1; Physical Inactivity; Sedentary Behavior; Gender Discrimination
Keywords: Mental health; Physical activity; Sedentary behavior; Gender equity
MeSH Terms: conditions — Sedentary Behavior; Sexism; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Uni4Move to sit less and move more — Co-create and implement an action plan to move more and sit less in the university context

SUMMARY:
Mental health, understood as the individual or group well-being at an emotional, psychological, and/or social level, affects up to 35% of university students, of whom only 16.4% seek or receive help from healthcare professionals. Despite this prevalence and its impact on academic performance and the challenges faced by universities in terms of limited resources to address this situation, most research tends to focus on primary and/or secondary education stages. Consequently, there is limited research on the reasons why university students experience mental health problems and why they do not seek help.

Physical activity and reducing sedentary behaviour could be protective factors for mental health in both children and adolescents. In this regard, according to data from the DESK-Uni at UVic-UCC, university students report engaging in low levels of physical activity, with female students reporting lower levels than male students. Additionally, adolescent girls report more mental health problems than boys. Therefore, there is a need for research and projects that consider the gender bias in health that exists in our society, including universities. This bias could explain why girls engage in less physical activity or claim to do so and why they experience more mental health problems. Thus, the purpose of the project is to improve or reduce gender inequalities within the university community and their impact on health behaviour (physical activity/sedentary behaviour) and mental health of both students and staff members.

Overall, the project aims to decrease the risks of experiencing mental health problems in the university environment by enhancing identification and promoting health-related behaviours that act as protective factors (e.g., physical activity). This will be done by considering the intersectionality of inequality axes present in our society and reproduced within the university setting. To do it, the Sustainable Development Goals (SDG; 3-4-5) will be taken in consideration.

DETAILED DESCRIPTION:
The university environment is not separate from society, which has experienced an increase in the prevalence of mental health problems following the COVID-19 pandemic. Similarly, the university environment is not immune to the gender biases of our society: in fact, the university itself could help perpetuate and reproduce these biases if not addressed. Therefore, it is necessary to investigate which social factors, such as gender construction, can influence aspects of health (mental health problems) and behaviour (engagement in physical activity or sedentary behaviour) within the university community.

Generally, the data provided by the university community are self-reported, often estimating levels of physical activity. Consequently, these low levels of physical activity may be even higher. Therefore, it is necessary to explore physical activity levels and sedentary behaviour using accelerometers and qualitatively examine, from a gender perspective, the reasons, barriers, and facilitators that influence engagement in physical activity and the improvement of sedentary behaviour among the university community.

On the other hand, while it is true that the UManresa university offers free psychological assistance to students (up to three visits per year), the understanding of mental health by the university community can affect the utilization of this service. For example, in a society that demands strength from "men," they may be more resistant to acknowledging their mental health problems, considering it a sign of weakness, and seeking help. Therefore, understanding how the university community perceives and interprets mental health is important: how it socially constructs the meaning of mental health problems and the role that gender plays in this construction.

In the face of this situation, the following questions arise: Is there a correlation between levels of physical activity, sedentary behaviour, and the mental health status of the university community? What social and gender factors in the university environment can lead to lower levels of physical activity and more mental health problems? What actions can the university community take to improve the current situation regarding health behaviours and mental health of the university community? Additionally, considering that levels of physical activity are influenced by gender inequity and that mental health problems are partly influenced by physical activity and sedentary behaviour, it is necessary to study the relationship between mental health, health behaviours, and gender perspective.

In fact, the report "Gender perspective in research at the University" (2017), coordinated by Tània Verge Mestre (Universitat Pompeu Fabra) and Teresa Cabruja Ubach (Universitat de Girona), found that the effective incorporation of a gender perspective in university teaching remained a pending challenge, despite the existing European regulatory framework. Therefore, social inequalities may continue to persist and reproduce within the university setting. In this sense, this project aims to incorporate a gender perspective to improve the quality of teaching and the social relevance of knowledge, technologies, and innovations (re)produced. Firstly, this perspective aims to improve mental health through levels of physical activity and sedentary behaviour in the university community, both of which are associated with gender biases. On the other hand, it aims to provide students with new tools to identify gender stereotypes, norms and roles to contribute to their critical thinking and acquire competencies that will enable them to avoid gender blindness in their future professional practice. Likewise, the gender perspective allows faculty and all university staff to pay attention to gender dynamics within the learning environment and take measures to ensure that the diversity of students is addressed, thereby impacting the mental health and potential health behaviours of the entire community.

Furthermore, it is necessary to explore both physical activity and sedentary behaviour using accelerometers and how these levels are linked to mental health problems and social determinants that influence the adoption or non-adoption of a healthy lifestyle and the social construction of gender and mental illness. Secondly, it is important to collaboratively develop an action plan among all stakeholders at the university level to implement the research project's findings. Finally, the action plan should be implemented from a gender perspective to reduce sedentary behaviour, improve levels of physical activity, and consequently reduce mental health problems. The results should be evaluated annually throughout the entire trajectory of the students.

The overall objective of the project is to co-create and implement an action plan at the university level from a gender perspective to improve levels of physical activity, reduce sedentary behaviour, and consequently decrease the risk of mental health problems among members of the university community.

The specific objectives include:

* Explore the acceptability and feasibility of implementing an action plan at the university level among different stakeholders from a gender perspective.
* Determine the levels of physical activity and sedentary behaviour among the university community and their correlation with mental health problems.
* Explore the experiences and factors (i.e gender inequity) that may influence the engagement in physical activity and sedentary behaviour, as well as the perception of mental health, among the university community.
* Create a gender-inclusive guide for university teaching that addresses the needs for improving levels of physical activity, reducing sedentary behaviour, and addressing mental health problems within the university community.

Each of the specific objectives will help confirm or refute the hypothesis posed. Broadly speaking, they can be categorized into two distinct types: those focusing on quantitative and biological outcomes (correlation between physical activity, sedentary behaviour, and mental health problems) and those interpreting, applying, or seeking to transfer the results through changes and actions in the daily life of the university community.

The study follows a mixed-methods approach using a Cooperative Planning Process (CPP) model. The CPP is a participatory approach that helps create dynamic social spaces to improve change processes in healthcare and health promotion in a fair and equitable manner. Additionally, participatory interventions aim to increase the fit (adaptation) of programs within the real-life contexts of the individuals involved (university community). In this sense, the CPP has been frequently used in promoting physical activity over the past decades. The CPP is a participatory intervention strategy that brings together stakeholders involved in the change process through egalitarian decision-making to plan, develop, and implement programs that align with the demands and needs of the target population. Therefore, the CPP addresses essential principles for interventions such as the multi-dimensionality of interventions (socioecological perspective), context-specific interventions (action plan), and the reciprocal adjustment between science and clinical practice.

To carry out the CPP, the project will be divided into different phases: i) Identification of the target population members and the needs of the stakeholders. ii) Development of an action plan to address the identified needs, including co-creation of the action plan for promoting physical activity, reducing sedentary behaviour, and raising awareness of mental health within the university community. iii) Establishing the feasibility and acceptability of the co-created action plan and adapting it based on the emerging needs through an initial application within the university community. iv) Implementation of the action plan through close collaboration with the target population and stakeholders. v) Evaluation of the success of the action plan and making necessary adaptations to ensure long-term sustainability.

By following this approach, the study aims to actively involve the university community and stakeholders in the planning, development, and implementation of interventions, ultimately promoting sustainable changes in physical activity, sedentary behaviour, and mental health throughout a gender perspective.

ELIGIBILITY:
Inclusion Criteria:

* Individuals involved in the university community, including students and staff members.
* No contraindication for participating in physical activity.

Exclusion Criteria:

* Lack of a B2 proficiency level in either Catalan or Spanish language (as determined by an official exam).
* Failure to provide informed consent to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will consist of healthy individuals from the university community who have no contraindications for engaging in physical activity and have no difficulties in understanding Spanish or Catalan.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-09-04 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Warwick-Edinburgh Mental Wellbeing Scales - WEMWBS at 2 years | Change from baseline at 2 years
  The 14-item scale WEMWBS has 5 response categories, summed to provide a single score. The items are all worded positively and cover both feeling and functioning aspects of mental wellbeing, thereby making the concept more accessible. At individual level 'minimum detectable change' has been calculated using different recommended methods giving results of 3 and 8 points. A change of 3 points means that scores on three items have improved or worsened by 1 point, or scores on one item have improved or worsened by 3 points. This suggests that the lower threshold of 3 points can be taken to represent 'meaningful change' between measurement points in individuals.

SECONDARY OUTCOMES:
Physical Activity Levels | Seven days a year during four years
  Levels of light, medium and vigorous physical activity weekly in minutes
Sedentary behavior time | Seven days a year during four years
  Number of total time in minutes of sedentary behavior
Sedentary behavior breaks | Seven days a year during four years
  Number of breaks (sit-to-stand transitions)
Sedentary behavior bouts | Seven days a year during four years
  Duration of bouts in minutes (>30, 30-60, <60).

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Jabardo Camprubí, PhD, Principal Investigator — Faculty of Health Science at Manresa
Locations (1):
- University of Vic-Central University of Catalunya, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the results of the study throughout posters, oral communications, webinars and publications in cientific journals
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Results will be share once a year
Access Criteria: Through out posters, communications, webinars and publications

REFERENCES:
- [Background] Bruffaerts R, Mortier P, Kiekens G, Auerbach RP, Cuijpers P, Demyttenaere K, Green JG, Nock MK, Kessler RC. Mental health problems in college freshmen: Prevalence and academic functioning. J Affect Disord. 2018 Jan 1;225:97-103. doi: 10.1016/j.jad.2017.07.044. Epub 2017 Jul 25. PMID 28802728
- [Background] Smith PJ, Merwin RM. The Role of Exercise in Management of Mental Health Disorders: An Integrative Review. Annu Rev Med. 2021 Jan 27;72:45-62. doi: 10.1146/annurev-med-060619-022943. Epub 2020 Nov 30. PMID 33256493
- [Background] Schuch FB, Vancampfort D. Physical activity, exercise, and mental disorders: it is time to move on. Trends Psychiatry Psychother. 2021 Jul-Sep;43(3):177-184. doi: 10.47626/2237-6089-2021-0237. Epub 2021 Apr 21. PMID 33890431